CLINICAL TRIAL: NCT00470444
Title: Transfusion Triggers in Cardiac Surgery
Acronym: TTRICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Blood Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 06-185
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2008-11

CONDITIONS: Cardiac Surgery
Keywords: Cardiac Surgery; Transfusion Medicine; Cardiac Anesthesia Risk Evaluation (CARE) Score of 3 or 4; (Dupuis J-Y et al, Anesthesiology 2001;94: 194-204)
MeSH Terms: interventions — Blood Transfusion; Erythrocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Liberal transfusion strategy
  Interventions: Procedure: Transfusion with Red Blood Cells; Biological: 1 unit of donated red blood cells
- 2 (Active Comparator): Restrictive transfusion strategy
  Interventions: Biological: 1 unit of donated red blood cells

INTERVENTIONS:
Procedure: Transfusion with Red Blood Cells — Units of donated Red blood cells
  Arms: 1
Biological: 1 unit of donated red blood cells — Units of red blood cells
  Arms: 1
Biological: 1 unit of donated red blood cells — Units of donated red blood cells
  Arms: 2

SUMMARY:
A high proportion of patients having cardiac surgery receive red cell transfusions. Yet, the investigators do not know whether transfusions are beneficial and they may be associated with harm. It is thus important to determine when a transfusion is required. The investigators will conduct a small pilot study at St. Michael's Hospital to address this issue. Patients having cardiac surgery will be allocated to one of two transfusion strategies with endpoints being compliance with the transfusion strategy and clinical outcome. The results of this study will be used to design a large definitive multicentered trial of these two transfusion strategies.

DETAILED DESCRIPTION:
The optimal hemoglobin concentrations for transfusion in the perioperative setting in patients having cardiac surgery have not been established, and red cell transfusion rates for these patients are high. In a recent retrospective study of seven Canadian centres, which included 11,812 cardiac surgical patients, 44% of patients received one or more red cell units, and the range of patients transfused was 28% to 60%. As morbidity and mortality may be dependent on the severity of anemia and administration of transfusions, it is essential to determine at what hemoglobin concentration physicians should be transfusing these patients, particularly because the efficacy of transfusion has not been established. However, as any definitive trial will require thousands of patients, and as there is variability in transfusion practices, preliminary studies need to be completed to ensure the feasibility of adherence to proposed transfusion strategies. This pilot study is the first of two pilot trials designed to address the question of optimum hemoglobin concentrations for transfusion in patients having cardiac surgery prior to undertaking a definitive randomized controlled trial. The purpose of this study is to determine adherence to transfusion strategies.

ELIGIBILITY:
Inclusion Criteria:

* Care Score of 3/4 or age >/= 80
* Signed informed consent

Exclusion Criteria:

* Patients who refuse participation
* Unable to or refuse blood products
* Involved in an autologous pre-donation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Overall adherence to the transfusion strategies defined as adherence to the transfusion strategies in 90% of patients in more than 90% of their days in hospital. | Day of surgery through to hospital discharge.

SECONDARY OUTCOMES:
1) enrollment rates 2) proportion of missing data 3) indicators for hypoxemia 4) mean number of red cell units used 5) clinical outcomes | Day of surgery through to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, MD, Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Dupuis JY, Wang F, Nathan H, Lam M, Grimes S, Bourke M. The cardiac anesthesia risk evaluation score: a clinically useful predictor of mortality and morbidity after cardiac surgery. Anesthesiology. 2001 Feb;94(2):194-204. doi: 10.1097/00000542-200102000-00006. PMID 11176081
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Shehata N, Burns LA, Nathan H, Hebert P, Hare GM, Fergusson D, Mazer CD. A randomized controlled pilot study of adherence to transfusion strategies in cardiac surgery. Transfusion. 2012 Jan;52(1):91-9. doi: 10.1111/j.1537-2995.2011.03236.x. Epub 2011 Jul 25. PMID 21790621